CLINICAL TRIAL: NCT05049213
Title: Investigating the Therapeutic Role of Topical Medical Treatment in Oral and Nasal Cavities on the Patients With Positive Severe Cute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Brief Title: Effect of Local Treatment(Carrageenan Nasal Spray and PVP-I Mouthwash) in Reducing Viral Load in Patients With COVID-19
Acronym: LT-COVID19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202106183RIND
Record Dates: First submitted 2021-09-16; First posted 2021-09-20 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Covid19; SARS-CoV 2 Infection
Keywords: COVID-19; Anti-septic; Carrageenan; Nasal spray; Povidone-Iodine(PVP-I); Gargle; Mouthwash
MeSH Terms: conditions — COVID-19 | interventions — Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Topical medical treatment (Experimental): Intranasal spray and oral gargling
  Interventions: Drug: Carrageenan nasal spray and 1% PVP- mouthwash and gargle

INTERVENTIONS:
Drug: Carrageenan nasal spray and 1% PVP- mouthwash and gargle — Day1 to Day7
  1. Intranasal spray 3 times/day, 2~3 spray/nostril/per time
  2. Oral gargling 3 times/day, 15cc/per time
  Other Names: BETADINE™ Cold Defense Nasal Spray and Povidone Iodine Mouthwash and Gargle

SUMMARY:
The goal of this study is to recruit confirmed Covid-19 patients, to evaluate whether the topical anti-septic can improve clinical outcome in early Severe acute respiratory syndrome coronavirus 2(SARS-CoV-2) infection. During the global pandemic period, an effective and highly available method once be identified, it will reduce the risk of disease transmission and lower the medical burden.

DETAILED DESCRIPTION:
Oral and nasal disinfection, a simple method with the application of commonly used antiseptic agents is frequently performed in the otolaryngology and dental practice. The ability to deactivate viral particles with a good safety profile may be an important benefit in the control of viral proliferation and shedding. Actually, multiple anti-septic agents demonstrated virucidal properties against SARS-CoV-2 in several in vitro studies. Among these, Povidone-Iodine (PVP-I), common usage in otolaryngology operation and topical therapy, showed high virucidal properties (0.45% PVP-I, throat spray, 4-log drop in viral load) and of great safety. There is also evidence that topical usage of saline can decrease the severity of upper respiratory tract infection. In addition, carrageenan, a sulphated polysaccharide purified from red marine algae, had shown efficacy in inhibiting multiple viruses, including in vitro studies of SARS-CoV-2. Some randomized controlled trials had also shown their abilities in improving patients' symptoms with a good safety profile. Multiple international organizations are conducting relating randomized clinical trials to evaluate whether the topical anti-septic improves clinical outcomes after early SARS-CoV-2 infection. The added value of topical antiseptic agents may be beneficial in improving symptoms, reducing viral load and alleviating the rate of disease progression. Due to relatively low risk, well-toleration to the general population, and highly available characteristics, the potential benefits of these agents deserve more attention.

The goal of this study is to investigate the changes in clinical symptoms and sequential laboratory data in confirmed COVID-19 adult patients at the early disease stage. By applying topical anti-septic which is frequently used in otolaryngology procedures, the investigators will evaluate the impact of this intervention on the symptoms, viral load and the rate of disease progression. During the global pandemic period, an effective and highly available method once be identified, it will reduce the risk of disease transmission and lower the medical burden.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 20 years of age
2. admission with a confirmed positive test for SARS-CoV-2 infection by reverse transcription polymerase chain reaction (RT- PCR)
3. disease onset (start of COVID-19 symptom and PCR test) for ≤ 120 hours
4. available informed consent of this study.
5. Full COVID-19 vaccination(at least after 2nd dose of TFDA-approved vaccine 14 days)

Exclusion Criteria:

1. receiving oxygen supply before intervention
2. known intolerance/allergy to the study drugs
3. pregnancy
4. sinus/oral operation within 30 days of the beginning of the study
5. using intranasal medication before randomization
6. no available informed consent
7. inability to self-care or reply to questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline naso-pharyngeal viral load quantified by RT-PCR at Day 8 | 7 days
  the mean change of viral titers of COVID-19 between Day 1 and Day 8 by RT-PCR test

SECONDARY OUTCOMES:
symptoms related to COVID-19 | 10 days
  including cough, fatigue, shortness of breath, loss of smell, hoarseness, chest pain, abdominal pain, diarrhea, headache, sore throat, muscle pain, etc and Quality of Life using the validated SinoNasal Outcome Tool-22 (SNOT-22, total score range 0-110, higher scores represent worse symptoms)
frequency of adverse effects of interest after anti-septic | 10 days
  including nasal discomfort, sneezing, epistaxis, headache and otalgia
number of days in an ICU | up to 14 days
  number of days in an ICU
number of days Non Invasive Ventilation (NIV) was required during hospitalization | up to 14 days
  NIV usage during hospitalization
mortality rates | up to 30 days
  mortality rates
length of hospitalization | up to 14 days
  length of hospitalization
days of discharge | up to 30 days
  free from quarantine

CONTACTS AND LOCATIONS:
Overall Officials: Te-Huei Yeh, MD-PhD, Principal Investigator — National Taiwan University Hospital, Department of Otolaryngology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
no plan to share individual participant data (IPD)

REFERENCES:
- [Result] Guenezan J, Garcia M, Strasters D, Jousselin C, Leveque N, Frasca D, Mimoz O. Povidone Iodine Mouthwash, Gargle, and Nasal Spray to Reduce Nasopharyngeal Viral Load in Patients With COVID-19: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Apr 1;147(4):400-401. doi: 10.1001/jamaoto.2020.5490. PMID 33538761
- [Result] Carrouel F, Valette M, Gadea E, Esparcieux A, Illes G, Langlois ME, Perrier H, Dussart C, Tramini P, Ribaud M, Bouscambert-Duchamp M, Bourgeois D. Use of an antiviral mouthwash as a barrier measure in the SARS-CoV-2 transmission in adults with asymptomatic to mild COVID-19: a multicentre, randomized, double-blind controlled trial. Clin Microbiol Infect. 2021 Oct;27(10):1494-1501. doi: 10.1016/j.cmi.2021.05.028. Epub 2021 May 24. PMID 34044151
- [Result] Hasan MJ, Rumi SKNF, Banu SS, Uddin AKMN, Islam MS, Arefin MK. Virucidal effect of povidone iodine on COVID-19 in the nasopharynx: A structured summary of a study protocol for an open-label randomized clinical trial. Trials. 2021 Jan 4;22(1):2. doi: 10.1186/s13063-020-04963-2. PMID 33397432